CLINICAL TRIAL: NCT00905229
Title: Comparing Different Routes and Doses of Phytonadione (Vitamin K) for Reversing Warfarin Treated Patients With Hip Fracture Before Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment problems
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: orit semana, haemek medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-09
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Bleeding; Complications
Keywords: hip fracture; warfarin; vitamin k; Phytonadione; INR level
MeSH Terms: conditions — Hemorrhage; Hip Fractures | interventions — Vitamin K 1; Vitamin K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PO (by mouth) (Active Comparator): 2.5 mg P.O Vitamin K
  Interventions: Drug: Phytonadione
- IV (intravenous ) (Active Comparator): 0.5 mg IV Vitamin K
  Interventions: Drug: Phytonadione

INTERVENTIONS:
Drug: Phytonadione — 2.5 mg po
  Other Names: vitamin k
  Arms: PO (by mouth)
Drug: Phytonadione — 0.5 mg IV
  Other Names: vitamin k
  Arms: IV (intravenous )

SUMMARY:
It is well known that femoral neck fractures carry a significant increase in patients' mortality and that surgical intervention is the preferred treatment.

Any delay in operating on such patients would inevitably increase their risk of developing complications. One of the reasons for such unintentional delay would be the hypercoagulative status of patients taking warfarin. The CHEST 2008 guidelines suggest reversing warfarin with Vitamin K for patients who need urgent operation. The aim of this study is to compare different roots and doses of Vitamin K.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture patients on warfarin

Exclusion Criteria:

* pregnancy
* vitamin k sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
International normalized ratio (INR) </= 1.2 | 3 days

SECONDARY OUTCOMES:
Bleeding | 6 weeks
Complications | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Background] Ansell J, Hirsh J, Hylek E, Jacobson A, Crowther M, Palareti G. Pharmacology and management of the vitamin K antagonists: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):160S-198S. doi: 10.1378/chest.08-0670. PMID 18574265
- [Background] Al-Rashid M, Parker MJ. Anticoagulation management in hip fracture patients on warfarin. Injury. 2005 Nov;36(11):1311-5. doi: 10.1016/j.injury.2005.05.004. PMID 16214475
- [Background] Lubetsky A, Yonath H, Olchovsky D, Loebstein R, Halkin H, Ezra D. Comparison of oral vs intravenous phytonadione (vitamin K1) in patients with excessive anticoagulation: a prospective randomized controlled study. Arch Intern Med. 2003 Nov 10;163(20):2469-73. doi: 10.1001/archinte.163.20.2469. PMID 14609783